CLINICAL TRIAL: NCT00950742
Title: Phase I Open Label Trial to Assess Safety of BIBW 2992 in Combination With Herceptin® in Patients With HER2-positive Advanced Breast Cancer.
Brief Title: Phase I Open Label Trial to Assess Safety of BIBW 2992 (Afatinib) in Combination With Herceptin® in Patients With HER2-positive Advanced Breast Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.68; 2009-010003-89 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Afatinib

ARMS (1):
- BIBW 2992 + Trastuzumab (Experimental): Find maximum tolerated dose of the non-marketed substance:BIBW 2992 given orally with fixed weekly infusion doses of 2mg/kg Herceptin. Escalating doses of BIBW 2992 starting at 20mg daily.
  Interventions: Drug: Trastuzumab; Drug: BIBW 2992

INTERVENTIONS:
Drug: Trastuzumab — Load: 4mg/kg-maintain:2mg/kg/week
Drug: BIBW 2992 — Increased dose cohorts from low dose to MTD

SUMMARY:
Study to determine the Maximum Tolerated dose of BIBW 2992 given in combination with Herceptin®

ELIGIBILITY:
Inclusion criteria:

1. Female patients aged >18 years.
2. Advanced or metastatic breast cancer that over-expresses HER2 (immunohistochemistry 3+ or 2+ and gene amplification by FISH). Prior treatment with Herceptin® or Lapatinib® (in the adjuvant or metastatic settings) is permitted but not required.

Exclusion criteria:

Patients with untreated or symptomatic brain metastases. Prior treatment with EGFR targeting therapies or treatment with EGFR- or HER2 inhibiting drugs within the past four weeks before the start of therapy or concomitantly with this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- United Kingdom (5):
  - 1200.68.44001 Boehringer Ingelheim Investigational Site, Brighton
  - 1200.68.44003 Boehringer Ingelheim Investigational Site, Cambridge
  - 1200.68.44005 Boehringer Ingelheim Investigational Site, Guildford
  - 1200.68.44004 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1200.68.44002 Boehringer Ingelheim Investigational Site, Truro

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label dose escalation study using a standard 3+3 dose escalation design, dose cohorts are presented here.
Groups:
- Afatinib 20mg + Herceptin: Patients received continuous daily dosing with Afatinib 20mg film-coated tablets and once weekly an intravenous infusion of Herceptin (4 mg/kg single loading dose to be followed by 2 mg/kg/week i.v.) until disease progression or lack of clinical benefit.
- Afatinib 30mg + Herceptin: Patients received continuous daily dosing with Afatinib 30mg film-coated tablets and once weekly an intravenous infusion of Herceptin (4 mg/kg single loading dose to be followed by 2 mg/kg/week i.v.) until disease progression or lack of clinical benefit.
Period: Overall Study
Arm/Group | Afatinib 20mg + Herceptin | Afatinib 30mg + Herceptin
Started | 16 (entered and treated) | 2 (entered and treated)
Completed | 0 | 0
Not Completed | 16 | 2
Not completed — Other Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Progressive Disease | 6 | 2
Not completed — Dose limiting toxicity | 6 | 0

BASELINE CHARACTERISTICS:
Population: Treated set
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 20mg + Herceptin | Afatinib 30mg + Herceptin | Total
Number analyzed (Participants) | 16 | 2 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.6) | 52.5 (6.4) | 61.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 2 | 18
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: Number of participants with DLT in the first cycle (28 days) for the determination of the maximum tolerated dose (MTD). Important Limitations and Caveats are provided in the respective section.
Time Frame: 28 days
Population: Treated set (TS). TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib. 3 patients were excluded as they were not evaluable for determination of maximum tolerated dose.
Measure: Number; unit: Participants
Groups:
- Afatinib 20mg + Herceptin: Patients received continuous daily dosing with Afatinib 20mg film-coated tablets and once weekly an intravenous infusion of Herceptin until disease progression or lack of clinical benefit. This group includes patients from the dose-escalation cohort and from the expansion cohort.
- Afatinib 30mg + Herceptin: Patients received continuous daily dosing with Afatinib 30mg film-coated tablets and once weekly an intravenous infusion of Herceptin until disease progression or lack of clinical benefit.
Arm/Group | Afatinib 20mg + Herceptin | Afatinib 30mg + Herceptin
Number analyzed (Participants) | 13 | 2
Participants | 4 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Afatinib in Combination With Herceptin(R)
Description: The MTD was defined as the highest dose at which no more than 1 of 6 patients experienced DLT. It was determined using a standard 3 + 3 dose escalation cohort design. To confirm the MTD, the MTD cohort was to be expanded to 18 patients with no more than 3/18 patients experiencing a DLT. Please refer to CAVEATs and Limitations.
Time Frame: 28 days
Population: TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib. 3 patients were excluded as they were not evaluable for determination of maximum tolerated dose.
Measure: Number; unit: mg
Groups:
- Afatinib: All patients received both Afatinib and Herceptin. Dose level 1 was continuous daily dosing with Afatinib 20mg tablets and once weekly an intravenous infusion of Herceptin. Dose level 2 was continuous daily dosing with Afatinib 30mg tablets and once weekly an intravenous infusion of Herceptin. Cycle length was 28 days.
Arm/Group | Afatinib
Number analyzed (Participants) | 8
mg | 20

3. Secondary Outcome: Number of Patients With Objective Response (OR)
Description: Objective tumor response based on response evaluation criteria in solid tumors (RECIST) version 1.1. OR is defined as complete response (CR) or partial response (PR).
Time Frame: Tumor assessment was performed at screening and every 2nd cycle until earliest time of progression, death or end of treatment.
Population: TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Measure: Number; unit: Participants
Arm/Group | Afatinib 20mg + Herceptin | Afatinib 30mg + Herceptin
Number analyzed (Participants) | 16 | 2
Participants | 2 | 0

4. Secondary Outcome: Number of Patients With Best Overall Response
Description: Best overall response based on response evaluation criteria in solid tumors (RECIST) version 1.1. Best overall response is defined as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) or not evaluable.
Time Frame: as for outcome 3
Population: TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Measure: Number; unit: Participants
Arm/Group | Afatinib 20mg + Herceptin | Afatinib 30mg + Herceptin
Number analyzed (Participants) | 16 | 2
Participants
  Complete Response | 0 | 0
  Partial Response | 2 | 0
  Stable Disease | 4 | 1
  Progressive Disease | 0 | 1
  Not evaluable | 10 | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as time from randomisation to disease progression or death whichever occurs first. Assessed by central independent review according to the response evaluation criteria in solid tumors (RECIST 1.1). Median time results from unstratified Kaplan-Meier estimates.
Time Frame: Baseline until disease progression, death or data cut-off.
Population: TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Afatinib 20mg + Herceptin | Afatinib 30mg + Herceptin
Number analyzed (Participants) | 16 | 2
Days | 113.0 [101.0 to 388.0] | 83.5 [56.0 to 111.0]

6. Secondary Outcome: Summary of Concentration of Afatinib in Plasma
Description: Pre-dose Concentrations of Afatinib in Plasma at Steady State on Days 8, 15 and 29 (Cpre,ss,8, Cpre,ss,15 and Cpre,ss,29) and Maximum Concentration of Afatinib in Plasma at Steady State (Cmax,ss).
Time Frame: 0.05 hours (h) before dosing and 0.5-1h, 2h, 3h, 4h, 5h, 6h, 8h after dosing
Population: Patients with no data available for the relevant parameter and dose were excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Afatinib 20mg + Herceptin: Patients received continuous daily dosing with Afatinib 20mg film-coated tablets and once weekly an intravenous infusion of Herceptin until disease progression or lack of clinical benefit.
Arm/Group | Afatinib 20mg + Herceptin
Number analyzed (Participants) | 16
ng/mL
  Cpre,ss,8 (N=11) | 9.75 (69.5)
  Cpre,ss,15 (N=13) | 9.94 (72.4)
  Cpre,ss,29 (N=8) | 9.15 (64.7)
  Cmax,ss (N=10) | 17.9 (80.9)

7. Secondary Outcome: Time From Dosing to the Maximum Concentration of Afatinib in Plasma at Steady State (Tmax,ss)
Description: tmax,ss represents the time from dosing to the maximum concentration of afatinib in plasma at steady state
Time Frame: 0.05 hours (h) before dosing and 0.5-1h, 2h, 3h, 4h, 5h, 6h, 8h after dosing
Population: Patients with no data available for the relevant parameter and dose were excluded from analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Afatinib 20mg + Herceptin
Number analyzed (Participants) | 11
hours | 4.25 [0.750 to 7.02]

8. Secondary Outcome: Summary of Concentration of Herceptin in Plasma
Description: Pre-dose Concentrations of Herceptin in Plasma on Days 8, 15 and 29 (Cpre,8, Cpre,15 and Cpre,29) and Maximum Concentration of Herceptin in Plasma on Days 1, 15 and 29 (Cmax,1, Cmax,15 and Cmax,29).
Time Frame: 0.05 hours (h) before dosing and 0.5-1h, 2h, 3h, 4h, 5h, 6h, 8h after dosing
Population: Patients with no data available for the relevant parameter and dose were excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 20mg + Herceptin
Number analyzed (Participants) | 16
ng/mL
  Cpre,8 (N=14) | 43600 (53.9)
  Cpre,15 (N=13) | 47200 (47.0)
  Cpre,29 (N=11) | 46200 (30.9)
  Cmax,1 (N=14) | 122000 (27.9)
  Cmax,15 (N=12) | 93000 (24.9)
  Cmax,29 (N=7) | 93200 (16.9)

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication (up to 1296 days)
Groups:
- Afatinib 20mg + Herceptin: Patients received continuous daily dosing with Afatinib 20mg film-coated tablets and once weekly an intravenous infusion of Herceptin (4 mg/kg single loading dose to be followed by 2 mg/kg/week i.v.) until disease progression.
- Afatinib 30mg + Herceptin: Patients received continuous daily dosing with Afatinib 30mg film-coated tablets and once weekly an intravenous infusion of Herceptin (4 mg/kg single loading dose to be followed by 2 mg/kg/week i.v.) until disease progression.
Arm/Group | Afatinib 20mg + Herceptin | Afatinib 30mg + Herceptin
Serious Adverse Events (participants affected / at risk) | 3/16 | 0/2
Other Adverse Events (participants affected / at risk) | 15/16 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 20mg + Herceptin (N=16) | Afatinib 30mg + Herceptin (N=2)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 20mg + Herceptin (N=16) | Afatinib 30mg + Herceptin (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 10 | 1
Oedema mouth (Gastrointestinal disorders) | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 6 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 1
Axillary pain (General disorders) | 1 | 0
Catheter site swelling (General disorders) | 1 | 0
Crepitations (General disorders) | 1 | 0
Fatigue (General disorders) | 9 | 1
Influenza like illness (General disorders) | 2 | 0
Local swelling (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Secretion discharge (General disorders) | 0 | 1
Spinal pain (General disorders) | 0 | 1
Tenderness (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Nail bed infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Purulent discharge (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ageusia (Nervous system disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Breast discharge (Reproductive system and breast disorders) | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 6 | 2
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
MTD was determined at 20mg afatinib when 1/6 pat. had DLT (3+3 design). Upon expansion of MTD cohort to 18 pat. recruitment was stopped when 4/13 pat. had DLT. No lower afatinib dose could be tested as 20mg was the lowest dose formulation available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.